CLINICAL TRIAL: NCT05767047
Title: A Phase 3, Multicenter, Open-label, Long-term Extension Study of Apremilast in Children 2 Years of Age or Older With Oral Ulcers Associated With Behçet's Disease or 5 Years of Age or Older With Juvenile Psoriatic Arthritis
Brief Title: A Study of Apremilast in Children With Oral Ulcers Associated With Behçet's Disease or Juvenile Psoriatic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190531; 2022-003024-41 (EudraCT Number); 2023-503433-21 (Other: EU CT number)
Record Dates: First submitted 2023-03-08; First posted 2023-03-14 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Behçet's Disease; Juvenile Psoriatic Arthritis
Keywords: Oral Ulcers; Behçet's Disease; Juvenile Psoriatic Arthritis; Apremilast; AMG 407; Otezla
MeSH Terms: conditions — Behcet Syndrome; Arthritis, Juvenile; Oral Ulcer | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apremilast (Experimental): Participants with a weight between ≥ 12 kg to < 20 kg will receive apremilast 10 mg BID (twice a day), participants with a weight between ≥ 20 kg to < 50 kg will receive 20 mg BID, and participants with a weight ≥ 50 kg will receive apremilast 30 mg BID.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Oral tablets or liquid suspension
  Other Names: AMG 407; Otezla; CC-10004

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of apremilast in subjects 2 years of age or older with oral ulcers associated with Behçets disease or 5 years of age or older with active juvenile psoriatic arthritis that have completed Study 20190530 or Study 20190529.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent / assent obtained
* Must have completed Week 52 on treatment on core study and must be < 18 years of age at the time the informed consent document is signed
* Age and sex specific body mass index (BMI) no lower in range than the 5th percentile on Centers for Disease Control (CDC growth chart) at enrollment
* Willing to adhere to study visit schedule and protocol requirements
* Must have acceptable benefit/risk for continued treatment with apremilast

Exclusion Criteria:

* Answer "yes" to any question on C-SSRS at Week 52 visit of core study
* Scheduled surgery or other interventions that would interrupt study participation
* Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment and for 30 days after last dose
* Female participants planning to become pregnant while on study through 30 days after last dose
* Female participants of childbearing potential with positive pregnancy test at Week 0
* Known sensitivity to any products to be administered during dosing

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2036-03-17 (Estimated); Study Completion 2036-03-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to approximately 4 years
  Adverse events will be classified using the Medical Dictionary for Regulatory Activities (MedDRA) classification system.
Columbia-Suicide Severity rating Scale (C-SSRS) | Up to approximately 4 years
  A questionnaire used to assess suicide risk.
Tanner Staging | Up to approximately 4 years
  Tanner Staging of sexual development assessment will be used to assess sexual maturity.
Change from Baseline in Body Weight | Up to approximately 4 years
Change from Baseline in Height | Up to approximately 4 years
Change from Baseline in Body Mass Index (BMI) | Up to approximately 4 years
Number of Participants with Clinically Significant Changes in Vital Signs | Up to approximately 4 years
Number of Participants with Clinically Significant Changes in Laboratory Parameters | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- General Hospital of Thessaloniki Ippokrateio, Thessaloniki, Greece
- Meir Medical Center, Kfar Saba, Israel
- Spain (2):
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Umraniye Egitim ve Arastirma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com